CLINICAL TRIAL: NCT07204431
Title: Efficacy of Respiratory Physiotherapy Treatment in Patients With Chronic Obstructive Disease in Elderly Patients.
Brief Title: Efficacy of Respiratory Physiotherapy Treatment in Chronic Obstructive Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, PhD. Physiotherapy, Universidad Pontificia de Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 092025
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: diaphragmatic expiratory exercises.; physiotherapy tecniques
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the PowerBreathe and PEP Therosold tools group. (Experimental)
  Interventions: Device: the PowerBreathe and PEP Therosold tools group.
- perform diaphragmatic breathing and expiratory exercises group. (Active Comparator)
  Interventions: Device: the PowerBreathe and PEP Therosold tools group.

INTERVENTIONS:
Device: the PowerBreathe and PEP Therosold tools group. — Initially, the following data were collected from each subject in addition to basic epidemiological data.

SUMMARY:
To test the effectiveness of a respiratory physiotherapy treatment plan in patients who have been diagnosed with chronic obstructive pulmonary disease, comparing with two randomized groups, for the performance of different respiratory musculature training protocols. Objectify the data obtained through ultrasound and spirometry, observing the differences obtained at the beginning and end of the study, verifying the efficacy of the PowerBreathe® and Therosold PEP® tools and the effectiveness of diaphragmatic, abdominal and expiratory exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic obstructive disease.
* Patients older than 65 years.
* Patients under age.
* Patients with cognitive ability to perform spirometry.
* Patients with physical ability to perform spirometry.

Exclusion Criteria:

* Patients without functional limitations in the respiratory system.
* Patients under 65 years of age.
* Patients with no cognitive ability to perform spirometry.
* Patients without physical ability to perform spirometry.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
peak inspiratory pressure (PIM). | 1 month.
  0 miminum ,200 maximum.
peak expiratory pressure. | 1 month.
  0 miminum ,200 maximum.
forced vital capacity. | 1 month.
  0 miminum ,200 maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pontificia de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Result] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Result] Lazzeri M, Lanza A, Bellini R, Bellofiore A, Cecchetto S, Colombo A, D'Abrosca F, Del Monaco C, Gaudiello G, Paneroni M, Privitera E, Retucci M, Rossi V, Santambrogio M, Sommariva M, Frigerio P. Respiratory physiotherapy in patients with COVID-19 infection in acute setting: a Position Paper of the Italian Association of Respiratory Physiotherapists (ARIR). Monaldi Arch Chest Dis. 2020 Mar 26;90(1). doi: 10.4081/monaldi.2020.1285. PMID 32236089
- [Result] Sanchez Mila Z, Rodriguez Sanz D, Martin Nieto A, Jimenez Lobo A, Ramos Hernandez M, Campon Chekroun A, Frutos Llanes R, Barragan Casas JM, Velazquez Saornil J. Effects of a respiratory and neurological rehabilitation treatment plan in post Covid-19 affected university students. Randomized clinical study. Chron Respir Dis. 2024 Jan-Dec;21:14799731241255967. doi: 10.1177/14799731241255967. PMID 38752418